CLINICAL TRIAL: NCT06126172
Title: Radiomics of Treatment-naive Prostate Cancer Patients on Multiparametric MRI for Risk Stratification and Treatment Outcomes Predictions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li-Jen Wang, Medical Imaging Department Director, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202002364B0
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Multiparametric MRI; Radiomics; Risk stratification; Recurrence; Prediction
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiparametric magnetic resonance imaging (Experimental): Detecting and localizing prostate cancers. The radiomics provide comprehensive quantitative information of all tumor data which could be used for risk stratification and prognosis prediction.
  Interventions: Diagnostic Test: Multiparametric magnetic resonance imaging (mpMRI)

INTERVENTIONS:
Diagnostic Test: Multiparametric magnetic resonance imaging (mpMRI) — Detecting and localizing prostate cancers and using radiomics extracted from prostate mpMRI for risk stratification patients of histological aggressiveness as well as to predict very early recurrence of PCA patients within 6 months after radical prostatectomy.

SUMMARY:
Prostate cancers (PCA) are a heterogeneous group which include indolent tumors that has no clinical significance to very aggressive cancer that could result in morbidities and mortality. Thus, an accurate risk stratification at the time of PCA diagnosis is crucial. The histological examination of PCA biopsy specimens could not accurately predict the final tumor aggressiveness shown on radical prostatectomy specimens because of heterogeneous distributions of the most malignant tumor cells. Prostate multiparametric magnetic resonance imaging (mpMRI) has been generally accepted to be the best imaging modality for detecting and localizing prostate cancers themselves. Furthermore, the rapid development of radiomics provide comprehensive quantitative information of all tumor data which could be used for risk stratification and prognosis prediction. Thus, this study plans to enroll 200 eligible patients who undergo prostate mpMRI first, followed by radical prostatectomy for prostate cancers. We use radiomics extracted from prostate mpMRI for risk stratification patients of histological aggressiveness as well as to predict very early recurrence of PCA patients within 6 months after radical prostatectomy.

DETAILED DESCRIPTION:
Prostate cancer is the 2nd most common malignancy in the world as well as the leading cancer in male population in Taiwan. The treatment selections of prostate cancer are limited by the uncertainty of its aggressiveness (i.e.: histological graded) and staging before treatment. Although prostate mpMRI has much better ability for detection and localization of prostate cancers than other imaging modalities and diagnostic tests, there is still gap for risk stratifications and treatment selection based on prostate mpMRI findings. Thus, a robust radiomics prediction models based on imaging biomarkers on prostate mpMRI with high prediction accuracy could fill the gap of misclassification of risk stratifications of prostate cancers, guides treatment selections and providing monitoring schedules for treated patients as well as early timely additional treatments (i.e.: target therapy or immunotherapy) for patients with high risk of early recurrence. Furthermore, radiomics could provide consistent information which help in decreasing interobserver and intra-observer variability of interpretating prostate cancer even in the use of PIRADS. In this way, this would save the fee of inappropriate or ineffective treatment and avoid unnecessary time and cost of monitoring low risk patients as well as improve patients' survivals and possibly life-quality as well.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 20 years old.
2. Suspected or confirmed prostate cancer.
3. Undergoing prostate mpMRI before clinical treatment.
4. Normal renal function(i.e.: estimated GFR ≧60).
5. No allergy history to gadolinium based contrast agent.
6. Agree to participate this study and sign informed consent.

Exclusion Criteria:

1. mpMRI photography not completed.
2. mpMRI images are damaged or poor in quality and cannot be interpreted.
3. Without pathological examination confirmed prostate cancer.
4. Patient withdraw informed consent.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MR characteristics assessment-T2WI | 1.5 year
  T2-weighted images (T2WI)
MR characteristics assessment- DWI | 1.5 year
  Axial diffusion weighted images (DWI)
MR characteristics assessment- ADC | 1.5 year
  Apparent diffusion coefficient maps (ADC)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jen Wang, M.D., M.P.H., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Li-Jen Wang, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Plan to make individual participant data.